CLINICAL TRIAL: NCT02297243
Title: The Sinopsys Lacrimal Stent Indicated for Sinus Irrigation Via Transcaruncular Ethmoid Sinus Access in Patients With Moderate to Severe Chronic Rhinosinusitis With Ethmoid Sinus Involvement
Brief Title: Sinopsys Lacrimal Stent Indicated for Sinus Irrigation
Acronym: SLS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sinopsys Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLS-US-02
Record Dates: First submitted 2014-11-14; First posted 2014-11-21 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Ethmoid Sinusitis
MeSH Terms: conditions — Ethmoid Sinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sinopsys Lacrimal Stent (Experimental): The Sinopsys Lacrimal Stent is indicated for use to create a transcaruncular ethmoid sinus access.
  Interventions: Device: Sinopsys Lacrimal Stent

INTERVENTIONS:
Device: Sinopsys Lacrimal Stent — The Sinopsys Lacrimal Stent is indicated for use to create a transcaruncular ethmoid sinus access.
  Other Names: SLS

SUMMARY:
The purpose of this study is to collect preliminary clinical data related to the safety and performance of the Sinopsys Lacrimal Stent.

DETAILED DESCRIPTION:
For purposes of this clinical study, the Sinopsys Lacrimal Stent is intended to provide a means of administering saline sinus irrigation via a transcaruncular-ethmoid sinus access in patients with moderate to severe chronic rhinosinusitis with ethmoid involvement. The purpose of the administration of saline irrigation is to reduce the intensity of symptoms of chronic rhinosinusitis in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. The Investigator has determined that the potential study subject has moderate to severe chronic rhinosinusitis with ethmoid involvement and has followed at least twelve (12) weeks of appropriate medical therapy prior to enrollment
2. Age ≥ 22 years
3. The potential study subject meets the American Academy of Otolaryngology - Head and Neck Surgery (AAO-HNS) criteria for chronic rhinosinusitis 12 weeks or longer of two or more of the following signs and symptoms:

   * Mucopurulent drainage (anterior, posterior, or both)
   * Nasal obstruction (congestion)
   * Facial pain-pressure-fullness, or
   * Decreased sense of smell

   AND inflammation is documented by one or more of the following findings:
   * Purulent (not clear) mucus or edema in the middle meatus or ethmoid region
   * Polyps in nasal cavity or the middle meatus, and/or
   * Radiographic imaging showing inﬂammation of the paranasal sinuses
4. SNOT-20 total score ≥ 41
5. CT scan (coronal view) confirms inflammation / involvement of the ethmoid sinuses
6. CT scan (coronal view) confirms depth of olfactory fossa is Keros classification 1 or 2.

Exclusion Criteria:

1. Sinus opacification score of ≤ 8 or ≥ 18 measured using the CT derived Lund -- Mackay scoring system
2. Isolated sinus disease evident on CT scan that would be unlikely to respond to target ethmoid treatment (e.g., isolated sphenoid or frontal disease)
3. Severe polyposis defined as Grade III or Grade IV polyposis using the adapted scale from Meltzer, 2006.
4. Prior ocular and/or sinus surgery for CRS
5. CT scan (coronal view) shows depth of olfactory fossa is Keros classification 3.
6. Prior surgical history, physical exam, nasal endoscopy and/or imaging studies suggest significant distortion of the craniofacial anatomy thus prohibiting adequate placement of the SLS
7. Presence of a sinonasal encepholocele as determined by CT scan
8. Presence of active HEENT infection including acute dacryocystitis
9. Febrile illness within 2 weeks and/or active pus from nose
10. Any sign of active ophthalmic disease, infection, or inflammation including the presence of severe ocular surface inflammatory disease or signs and symptoms of "dry eye disease" as determined by physical exam which could be exacerbated by the presence of the device
11. Current use of topical medications for the eye to treat an active ophthalmic disease
12. HbA1c level of ≥ 7.5% at the time of screening, current chemotherapy, or other immune compromised conditions

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
SNOT - 20 | 18 Weeks
  Chronic Rhinosinusitis symptoms as measured by SNOT-20 scores from baseline to 18 weeks follow-up (1, 4, 8, 12, and 18)
Patency will be confirmed post procedure with passive flow through the SLS lumen by instilling 2-4 drops of sterile saline into the stented medial fornix and observing drainage. | 18 Weeks
  Patients will be trained for self-administration of saline irrigation prior to the discharge home. Subjects will be instructed how to observe for stent patency and to report problems with flow to the Investigator.
Safety: Incidence and occurrence of anticipated and unanticipated adverse events | 18 Weeks
  Assessment of the incidence and occurrence of anticipated and unanticipated adverse events reported during the 18 weeks of the clinical study.

SECONDARY OUTCOMES:
Lund-MacKay CT Scores | 12 Weeks
  Comparison of baseline and 12 weeks
Lund-Kennedy Nasal Endoscopy Scores | 12 Weeks
  Comparison of baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Teena Augustino, Study Director — Sinopsys Surgical Inc.
Locations (3):
- United States (3):
  - Stanford University, Stanford, California
  - Front Range ENT, Greeley, Colorado
  - Advanced ENT and Allergy, Louisville, Kentucky